CLINICAL TRIAL: NCT03696628
Title: Modeling and Pharmacological Targeting of Genetic Cardiomyopathy in Children Via Cardiomyocytes Derived From Induced Pluripotent Stem Cells
Brief Title: Modeling and Pharmacological Targeting of Genetic Cardiomyopathy in Children Via Cardiomyocytes Derived From Induced Pluripotent Stem Cells (DMDstem)
Acronym: DMDstem
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 9806; 2017-A01589-44 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2018-08-07; First posted 2018-10-04 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-07

CONDITIONS: Cardiomyopathy, Familial
Keywords: Cardiomyocytes; Induced pluripotent stem cells; Genetic cardiomyopathy
MeSH Terms: conditions — Cardiomyopathies | interventions — Restraint, Physical; Hematologic Tests

STUDY DESIGN:
Intervention Model Description: All participants receive the same intervention throughout the protocol, no matter if they are "healthy children" or "cardiomyopathic children".
Masking Description: Open : no masking us used. All involved know the identity of the intervention assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy children (Other): Blood test with generated hiPSC-cardiomyocytes Physical Examination. Electrocardiogram. Echocardiography.
  Interventions: Other: Electrocardiogram; Other: physical examination; Other: echocardiography; Biological: blood test
- Cardiomyopathic children (Other): Blood test with generated hiPSC-cardiomyocytes Physical Examination. Electrocardiogram. Echocardiography.
  Interventions: Other: Electrocardiogram; Other: physical examination; Other: echocardiography; Biological: blood test

INTERVENTIONS:
Other: Electrocardiogram — heart testing
Other: physical examination — done by the investigator
Other: echocardiography — heart testing
Biological: blood test — A sample of blood will be taken to each patient or healthy children in order to generate hiPSC-cardiomyocytes

SUMMARY:
Interventional, cross-sectional biomedical study of children with genetic cardiomyopathy and healthy children. The aim is to generate, via induced human pluripotent stem cells (hiPSC), "patient-specific" cardiomyocytes (CMs) (hiPSC-CMs) to study the molecular mechanisms of cardiomyopathies of genetic origin.

DETAILED DESCRIPTION:
Interventional, cross-sectional biomedical study of children with genetic cardiomyopathy and healthy children. The aim is to generate, via induced human pluripotent stem cells (hiPSC), "patient-specific" cardiomyocytes (CMs) (hiPSC-CMs) to study the molecular mechanisms of cardiomyopathies of genetic origin.

The study will be proposed to the parents or legal guardians of the children from 0 to 17 included sent in pediatric cardiology consultation to the University Hospital of Montpellier as part of their usual follow-up or a health check (control) .

The only direct intervention performed on the patient is a venous blood sample. The volume of blood collected will be lower than the thresholds defined in the Decree of December 2nd, 2016 on minimal risks in biomedical research (3 ml).

ELIGIBILITY:
Group 1 : Child with genetic cardiomyopathy

Inclusion criteria

* Child from 0 to 17 years old included
* Bearer or at risk of cardiomyopathy of genetic origin. Written and informed consent of parents or guardians of legal guardians
* Affiliation or beneficiary of a social security scheme

Criterion of non-inclusion

. Cardiomyopathy of non-genetic origin (metabolic, toxic, malformative, etc.)

Group 2 : Healthy child

Inclusion criteria

* Children aged 0 to 17 years old
* Normal assessment: clinical examination, ECG, echocardiography
* Written and informed consent
* Affiliation or beneficiary of a social security scheme

Criterion of non-inclusion

* Heart, muscle or respiratory disease
* Treatment with cardiac resonance
* Other chronic diseases (diabetes, neuropathy, kidney failure, tumor)

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
hiPSC-cardiomyocytes culture | Inclusion visit
  Blood test with generated hiPSC-cardiomyocytes

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Arnaud de Villeneuve, Montpellier, Occitanie, France

REFERENCES:
- [Result] Souidi M, Amedro P, Meyer P, Desprat R, Lemaitre JM, Rivier F, Lacampagne A, Meli AC. Generation of three Duchenne Muscular Dystrophy patient-specific induced pluripotent stem cell lines DMD_YoTaz_PhyMedEXp, DMD_RaPer_PhyMedEXp, DMD_OuMen_PhyMedEXp (INSRMi008-A, INSRMi009-A and INSRMi010-A). Stem Cell Res. 2020 Dec;49:102094. doi: 10.1016/j.scr.2020.102094. Epub 2020 Nov 19. PMID 33246213